CLINICAL TRIAL: NCT00633581
Title: Efficacy of High Dose Vitamin C Parenteral Supplement on Amelioration of Fatigue in Company Workers After Work: A Double-Blind, Randomized Controlled Trial
Brief Title: Efficacy of Vitamin C Injection on Fatigue in Workers After Work
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: DongGuk University (Other)
Collaborators: Korean Association For Vitamin Research (Unknown)
Responsible Party: ChangHwan Yeom, Kwandong University College of Medicine Myungji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: DUIH 2008-1-1
Record Dates: First submitted 2008-03-03; First posted 2008-03-12 (Estimated); Last update posted 2009-04-10 (Estimated); Status verified 2009-04

CONDITIONS: Fatigue
Keywords: fatigue; ascorbic acid; oxidative stress
MeSH Terms: conditions — Fatigue | interventions — Ascorbic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Intravenous injections of 10 grams(20ml as a solution) of vitamin C with 100ml of normal saline over 30 minutes.
  Interventions: Dietary Supplement: Ascorbic acid (Vitamin C)
- 2 (Placebo Comparator): Intravenous injections of 120ml of normal saline over 30 minutes.
  Interventions: Dietary Supplement: Normal saline

INTERVENTIONS:
Dietary Supplement: Ascorbic acid (Vitamin C) — Single intravenous injection of vitamin C 10g(20ml) with 100ml of normal saline over 30 minutes
  Other Names: Ascorbic acid; Merit C
  Arms: 1
Dietary Supplement: Normal saline — Single intravenous injection of 120ml of normal saline over 30 minutes
  Arms: 2

SUMMARY:
Fatigue is one of the most frequently observed symptoms for company workers, and oxidative stress is regarded as one of its cause. Vitamin C is a well-known antioxidant, and the investigators seek for evidence of the efficacy of high dose vitamin C parenteral supplement on fatigue symptoms of company workers after work.

DETAILED DESCRIPTION:
Previous studies dealing with vitamin C were focusing on terminal cancer patients or those with chronic fatigue syndrome. Since used drug dosage and the ways of administering vitamin C were not identical, the results were not consistent throughout those studies. This study is aimed to evaluate the efficacy of high dose vitamin C with parenteral supplement on relieving fatigue for apparently healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Company workers working at least 5 days a week from morning to evening
* Volunteers who provided written informed consent

Exclusion Criteria:

* Acute illness
* Chronic disease such as diabetes, hypertension, liver disease, or renal disease
* Previous history of renal stone or gout
* Pregnant or lactating women
* Hypersensitivity to vitamins or intravenous injections
* History of vitamin supplements orally or parenterally within 2 days

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Degree of fatigue at the point of time with visual analogue scale from 0 to 10 | Before intravenous vitamin C injection and right after completing injections, and one day later

SECONDARY OUTCOMES:
Reactive oxygen species | Before intravenous vitamin C injections, right after completing injections, and one day later
Plasma vitamin C level | Before intravenous vitamin C injections and right after completing injections

CONTACTS AND LOCATIONS:
Overall Officials: Chang H Yeom, MD, PhD, Principal Investigator — KwanDong University Myungji Hospital
Locations (1):
- DongGuk University International Hospital, Goyang-si, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Bates DW, Schmitt W, Buchwald D, Ware NC, Lee J, Thoyer E, Kornish RJ, Komaroff AL. Prevalence of fatigue and chronic fatigue syndrome in a primary care practice. Arch Intern Med. 1993 Dec 27;153(24):2759-65. PMID 8257251
- [Background] Skapinakis P, Lewis G, Meltzer H. Clarifying the relationship between unexplained chronic fatigue and psychiatric morbidity: results from a community survey in Great Britain. Am J Psychiatry. 2000 Sep;157(9):1492-8. doi: 10.1176/appi.ajp.157.9.1492. PMID 10964867
- [Background] Logan AC. Nutritional strategies for treating chronic fatigue syndrome. Altern Med Rev. 2001 Feb;6(1):4-6. No abstract available. PMID 11207453
- [Background] Richards RS, Roberts TK, McGregor NR, Dunstan RH, Butt HL. Blood parameters indicative of oxidative stress are associated with symptom expression in chronic fatigue syndrome. Redox Rep. 2000;5(1):35-41. doi: 10.1179/rer.2000.5.1.35. PMID 10905542
- [Background] Cairns R, Hotopf M. A systematic review describing the prognosis of chronic fatigue syndrome. Occup Med (Lond). 2005 Jan;55(1):20-31. doi: 10.1093/occmed/kqi013. PMID 15699087
- [Background] Grossi G, Perski A, Evengard B, Blomkvist V, Orth-Gomer K. Physiological correlates of burnout among women. J Psychosom Res. 2003 Oct;55(4):309-16. doi: 10.1016/s0022-3999(02)00633-5. PMID 14507541
- [Background] Avalos I, Chung CP, Oeser A, Milne GL, Morrow JD, Gebretsadik T, Shintani A, Yu C, Stein CM. Oxidative stress in systemic lupus erythematosus: relationship to disease activity and symptoms. Lupus. 2007;16(3):195-200. doi: 10.1177/0961203306075802. PMID 17432105
- [Background] Powers SK, Hamilton K. Antioxidants and exercise. Clin Sports Med. 1999 Jul;18(3):525-36. doi: 10.1016/s0278-5919(05)70166-6. PMID 10410839
- [Background] Mantovani G, Maccio A, Madeddu C, Mura L, Massa E, Gramignano G, Lusso MR, Murgia V, Camboni P, Ferreli L. Reactive oxygen species, antioxidant mechanisms and serum cytokine levels in cancer patients: impact of an antioxidant treatment. J Cell Mol Med. 2002 Oct-Dec;6(4):570-82. doi: 10.1111/j.1582-4934.2002.tb00455.x. PMID 12611641
- [Background] Kennedy G, Spence VA, McLaren M, Hill A, Underwood C, Belch JJ. Oxidative stress levels are raised in chronic fatigue syndrome and are associated with clinical symptoms. Free Radic Biol Med. 2005 Sep 1;39(5):584-9. doi: 10.1016/j.freeradbiomed.2005.04.020. PMID 16085177
- [Background] Bryer SC, Goldfarb AH. Effect of high dose vitamin C supplementation on muscle soreness, damage, function, and oxidative stress to eccentric exercise. Int J Sport Nutr Exerc Metab. 2006 Jun;16(3):270-80. doi: 10.1123/ijsnem.16.3.270. PMID 16948483
- [Background] Sanchez-Moreno C, Cano MP, de Ancos B, Plaza L, Olmedilla B, Granado F, Martin A. Consumption of high-pressurized vegetable soup increases plasma vitamin C and decreases oxidative stress and inflammatory biomarkers in healthy humans. J Nutr. 2004 Nov;134(11):3021-5. doi: 10.1093/jn/134.11.3021. PMID 15514269
- [Background] Weijl NI, Elsendoorn TJ, Lentjes EG, Hopman GD, Wipkink-Bakker A, Zwinderman AH, Cleton FJ, Osanto S. Supplementation with antioxidant micronutrients and chemotherapy-induced toxicity in cancer patients treated with cisplatin-based chemotherapy: a randomised, double-blind, placebo-controlled study. Eur J Cancer. 2004 Jul;40(11):1713-23. doi: 10.1016/j.ejca.2004.02.029. PMID 15251161
- [Background] Mayland CR, Bennett MI, Allan K. Vitamin C deficiency in cancer patients. Palliat Med. 2005 Jan;19(1):17-20. doi: 10.1191/0269216305pm970oa. PMID 15690864
- [Background] Knekt P, Ritz J, Pereira MA, O'Reilly EJ, Augustsson K, Fraser GE, Goldbourt U, Heitmann BL, Hallmans G, Liu S, Pietinen P, Spiegelman D, Stevens J, Virtamo J, Willett WC, Rimm EB, Ascherio A. Antioxidant vitamins and coronary heart disease risk: a pooled analysis of 9 cohorts. Am J Clin Nutr. 2004 Dec;80(6):1508-20. doi: 10.1093/ajcn/80.6.1508. PMID 15585762
- [Derived] Suh SY, Bae WK, Ahn HY, Choi SE, Jung GC, Yeom CH. Intravenous vitamin C administration reduces fatigue in office workers: a double-blind randomized controlled trial. Nutr J. 2012 Jan 20;11:7. doi: 10.1186/1475-2891-11-7. PMID 22264303